CLINICAL TRIAL: NCT00518934
Title: Study for Safety and Efficiency of Therapeutic Angiogenesis for Patients With Limb Ischemia by Transplantation of Human Cord Blood Mononuclear Cell
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007-04-064
Record Dates: First submitted 2007-08-19; First posted 2007-08-21 (Estimated); Last update posted 2007-08-21 (Estimated); Status verified 2007-05

CONDITIONS: Ischemia
Keywords: Safety and efficiency of angiogenesis for patients with limb; ischemia by transplantation of human cord blood mononuclear; cells
MeSH Terms: conditions — Ischemia | interventions — Safety

INTERVENTIONS:
Other: Study for safety and efficiency of therapeutic angiogenesis for patients with limb ischemia by transplantation of human cord blood mononuclear cell

SUMMARY:
The purpose of this study is to analyze the safety and efficiency of therapeutic angiogenesis for patients with limb ischemia by transplantation of human cord blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:Patients with ischemic symptoms such as claudication, rest pain or nonhealing ischemic wound

* Without evidence of improvement in response to conventional medical therapy
* Not candidates for surgical intervention or radiologic intervention

Exclusion Criteria:

* Malignant disease
* More than 60 years old
* Other significant medical conditions, including diabetes mellitus, hypertension, hyperlipidemia, etc.

Max Age: 60 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ik Kim, Professor, Study Director — Professor of division of vascular surgery, Samsung Medical Center, Sungkyunkwan University of School of Medicine
Locations (1):
- Samsung Medical Center, Sungkyunkwan University School of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Kim DI, Kim MJ, Joh JH, Shin SW, Do YS, Moon JY, Kim NR, Lim JE, Kim AK, Eo HS, Kim BS, Cho SW, Yang SH, Park CJ, Shim JS. Angiogenesis facilitated by autologous whole bone marrow stem cell transplantation for Buerger's disease. Stem Cells. 2006 May;24(5):1194-200. doi: 10.1634/stemcells.2005-0349. Epub 2006 Jan 26. PMID 16439614